CLINICAL TRIAL: NCT06735599
Title: Effects of Wild Blueberry Consumption on Gut, Brain, and Cardiovascular Health in Non-Hispanic Black and White Adults With High Blood Pressure
Brief Title: Wild Blueberries for Gut, Brain, and Heart Health in Adults With High Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Rafaela G. Feresin, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H23563
Record Dates: First submitted 2024-11-05; First posted 2024-12-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hypertension (Without Type 2 Diabetes Mellitus); High Blood Pressure; Male; Female; Adult; Cognition; Endothelial Function (Reactive Hyperemia); Oxidative Stress; Diet; Overweight; Body Composition Measurement; Gut Microbiome; Arterial Stiffness; Caucasian Whites; Inflammation; Microvascular Function
Keywords: Blueberries; Hypertension; Overweight; High Blood Pressure; Endothelial Function; Cognitive Function; Dietary intervention; functional foods; gut microbiota; arterial stiffness; microvascular function
MeSH Terms: conditions — Hypertension; Hyperemia; Overweight; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wild Blueberry (Experimental): 22 g of freeze-dried wild blueberry freeze-dried powder per day
  Interventions: Dietary Supplement: Wild Blueberry
- Placebo (Placebo Comparator): 22 g of freeze-dried macronutrient-matched placebo powder per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wild Blueberry — Daily consumption of 22 g of freeze-dried wild blueberry freeze-dried powder for 8 weeks
  Arms: Wild Blueberry
Dietary Supplement: Placebo — Daily consumption of 22 g of freeze-dried macronutrient-matched placebo powder for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effectiveness of wild blueberries on cardiovascular health, cognitive function, and gut microbiota composition in non-Hispanic Black and White adults with elevated blood pressure.

DETAILED DESCRIPTION:
Hypertension (HTN), or high blood pressure (BP) is a major modifiable risk factor for heart disease, the leading cause of death worldwide. In the U.S., 121.5 million adults have high BP and only 25% have their BP under control. The 2022 Heart Disease and Stroke Statistics indicated that the incidence of high BP was higher among non-Hispanic Black (NHB) compared to non-Hispanic White (NHW) adults. Berries are rich in fiber and phytochemicals and have several health benefits. A 14-year follow-up of the Nurses' Health Study I and II and the Health Professional Follow-Up Study revealed a significant reduction in the risk of HTN (8%) among individuals in the highest quintile of anthocyanin intake compared to the lowest quintile. Blueberries are rich in fiber and phytochemicals that may be responsible for their health benefits. Studies have shown that daily blueberry consumption improves heart, cognitive, and intestinal health in different populations. Yet, a comprehensive study exploring and comparing the effectiveness of wild blueberries for cardiovascular, intestinal, and cognitive function parameters and their association in NHB and NHW adults with high BP has not been conducted to date.

Thus, the overall objective of this timely study is to determine and compare the effectiveness of a freeze-dried wild blueberry intervention on cardiovascular and gut health in NHB and NHW adults with high BP and assess whether these health benefits are associated with improvements in memory and other important thinking abilities for productivity and quality of life.

Therefore, this 8-week randomized, placebo-controlled parallel-arm clinical trial aims to assess whether daily consumption of 22 g of freeze-dried wild blueberry powder improves gut, cardiovascular, and cognitive function in NHB and NHW adults with elevated blood pressure and stage 1 hypertension. Investigators hypothesize that daily consumption of wild blueberries will improve cardiovascular parameters, gut dysbiosis, and cognitive function. To test these hypotheses, the following specific aims are proposed. To investigate whether daily consumption of 22 g of freeze-dried wild blueberry powder:

* Reduces BP, improves endothelial function, arterial stiffness, and microcirculation.
* Favorably modulates gut microbiota composition.
* Improves cognitive function (verbal memory and executive functions [inhibition, working memory, cognitive flexibility]).
* Improves serum markers of oxidative stress and inflammation.

Additionally, investigators will also explore whether changes in the gut microbiota are associated with changes in cardiometabolic and cognitive function outcomes and whether changes in cardiometabolic outcomes are associated with changes in cognitive function parameters globally and within each race.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 45-65 years of age
* Diagnosis of elevated blood pressure or stage 1 hypertension (systolic blood pressure = 120-139 mmHg and/or diastolic blood pressure = 80-89 mmHg) for at least 6 months
* BMI 25-30 kg/m2 via anthropometric measurements.
* Ability to give consent

Exclusion Criteria:

* Allergies to berries
* Use of one hypertensive drug for less than three months
* Use of more than one anti-hypertensive drug, insulin, antibiotics, and anti-inflammatory drugs, active cancer, gastrointestinal, renal, cardiovascular, thyroid, and neurological disorders or severe head injury
* Smoking
* Alcohol consumption (>2 drinks/day)
* Consuming antioxidant, probiotic, and prebiotic supplements
* Pregnant or lactating
* Participating in a weight loss program

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | Baseline, 4 weeks, and 8 weeks
  Assessment of whole-day ambulatory blood pressure during daytime and nighttime periods.
Pulse Wave Velocity | Baseline, 4 weeks, and 8 weeks
  Arterial Stiffness will be measured by pulse wave velocity using SphygmCor

SECONDARY OUTCOMES:
Reactive Hyperemia Index | Baseline, 4 weeks, and 8 weeks
  Assessment of endothelial function in response to increased shear stress using EndoPAT2000
Gut Microbiota Composition | Baseline, 4 weeks, and 8 weeks
  Analysis of stool sample for determination of absolute levels of bacteria and relative species composition
Global Cognitive Ability | Screening
  Measured using NIH Toolbox Picture Vocabulary and Oral Reading Recognition test
Performance Validity | Baseline, 4 weeks, and 8 weeks
  Assessed using Rey 15
Verbal Memory & Recognition | Baseline, 4 weeks, and 8 weeks
  Measured using Rey Auditory Verbal Learning Test with appropriate alternate forms
Cognitive Inhibition | Baseline, 4 weeks, and 8 weeks
  Assessed using Delis-Kaplan Executive Function System Trails and Verbal Fluency Switching
Working Memory | Baseline, 4 weeks, and 8 weeks
  Measured using Digit Span and NIH Toolbox List Sorting
Processing Speed | Baseline, 4 weeks, and 8 weeks
  Measured using NIH Toolbox Pattern Comparison and Oral Symbol Digit tests
Associative Memory | Baseline, 4 weeks, and 8 weeks
  Measured using NIH Toolbox Face Name Associative Memory Exam and Face Name Associative Memory Exam Delay tests
Attention | Baseline, 4 weeks, and 8 weeks
  Assessed using Wechsler Adult Intelligence Scale - IV and Rey Auditory Verbal Learning Test Trial 1.
Problem-Solving | Baseline, 4 weeks, and 8 weeks
  Assessed using NIH Toolbox Visual Reasoning

OTHER OUTCOMES:
Percent Maximal Microvascular Blood Flow | Baseline, 4 weeks, and 8 weeks
  Micro-vessel blood flow in response to local heating stimulus will be assessed using a Laser Doppler
Circulating Markers of Inflammation and Oxidative Stress | Baseline, 4 weeks, and 8 weeks
  Measurement of concentrations of circulating markers of inflammation such as CRP and oxidative stress such as TBARS in blood plasma and serum samples.
Urinary Polyphenolic Metabolites | Baseline, 4 weeks, and 8 weeks
  24-hour urine collection samples will be assessed for polyphenol metabolites
Body Fat | Baseline, 4 weeks, 8 weeks
  DEXA will be used to assess body fat mass

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela G Feresin, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krikorian R, Skelton MR, Summer SS, Shidler MD, Sullivan PG. Blueberry Supplementation in Midlife for Dementia Risk Reduction. Nutrients. 2022 Apr 13;14(8):1619. doi: 10.3390/nu14081619. PMID 35458181
- [Background] Johnson SA, Figueroa A, Navaei N, Wong A, Kalfon R, Ormsbee LT, Feresin RG, Elam ML, Hooshmand S, Payton ME, Arjmandi BH. Daily blueberry consumption improves blood pressure and arterial stiffness in postmenopausal women with pre- and stage 1-hypertension: a randomized, double-blind, placebo-controlled clinical trial. J Acad Nutr Diet. 2015 Mar;115(3):369-377. doi: 10.1016/j.jand.2014.11.001. Epub 2015 Jan 8. PMID 25578927
- [Background] Cassidy A, O'Reilly EJ, Kay C, Sampson L, Franz M, Forman JP, Curhan G, Rimm EB. Habitual intake of flavonoid subclasses and incident hypertension in adults. Am J Clin Nutr. 2011 Feb;93(2):338-47. doi: 10.3945/ajcn.110.006783. Epub 2010 Nov 24. PMID 21106916
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371